CLINICAL TRIAL: NCT01104103
Title: The BOA(R)-Constricting IV Band: A Single Blind, Cohort Study of Effectiveness
Brief Title: Effectiveness Study of the BOA(R)-Constricting IV Band
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pre-determined stopping point met with signficant difference between intervention and control groups.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: North American Rescue, LLC (Unknown)
Responsible Party: Principal Investigator, Richard Bradley, Associate Professor - Emergency Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NAR UTH 001
Record Dates: First submitted 2010-04-09; First posted 2010-04-15 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-07

CONDITIONS: Catheterization, Peripheral
Keywords: Catheterization, Peripheral; Disposable Equipment; Emergency Medical Technicians; Emergency Nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOA(R) (Experimental): Nurse or paramedic uses the BOA(R)-Constricting IV Band to attempt placement of an upper extremity IV in an adult
  Interventions: Device: BOA(R)-Constricting IV Band
- Standard care (Active Comparator): Nurse or paramedic uses standard IV starting technique in the upper extremity of adults
  Interventions: Device: Standard elastic constricting band

INTERVENTIONS:
Device: BOA(R)-Constricting IV Band — Device applied in accordance with manufacturer's instructions
  Other Names: NSN: 6515-01-537-2611
  Arms: BOA(R)
Device: Standard elastic constricting band — Standard therapy
  Other Names: elastic constricting band (Cardinal Health; McGaw Park, IL)
  Arms: Standard care

SUMMARY:
The purpose of this study is to determine whether the BOA(R)-Constricting IV Band is superior to standard methods for starting an IV.

DETAILED DESCRIPTION:
We will test the hypothesis that paramedics and nurses treating in- and out-of-hospital patients with a BOA(R)-Constricting IV Band, compared to paramedics using standard treatment, will have better success rates for peripheral IV access.

ELIGIBILITY:
Inclusion Criteria:

* Paramedics employed by the City of Houston or nurses employed by Memorial Hermann Hospital - Texas Medical Center
* Agree to participate through written consent process

Exclusion Criteria:

* City of Houston paramedics and Memorial Hermann Hospital - Texas Medical Center nurses who do not provide written informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard N Bradley, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Houston Fire Department, Houston, Texas
  - Memorial Hermann Hospital-Texas Medical Center, Houston, Texas

REFERENCES:
- [Background] Black KJ, Pusic MV, Harmidy D, McGillivray D. Pediatric intravenous insertion in the emergency department: bevel up or bevel down? Pediatr Emerg Care. 2005 Nov;21(11):707-11. doi: 10.1097/01.pec.0000186422.77140.1f. PMID 16280942
- [Background] Meier J, Schreier E. Human plasma levels of some anti-migraine drugs. Headache. 1976 Jul;16(3):96-104. doi: 10.1111/j.1526-4610.1976.hed1603096.x. No abstract available. PMID 965227
- [Background] Jacobson AF, Winslow EH. Variables influencing intravenous catheter insertion difficulty and failure: an analysis of 339 intravenous catheter insertions. Heart Lung. 2005 Sep-Oct;34(5):345-59. doi: 10.1016/j.hrtlng.2005.04.002. PMID 16157191
- [Background] Lapostolle F, Catineau J, Garrigue B, Monmarteau V, Houssaye T, Vecci I, Treoux V, Hospital B, Crocheton N, Adnet F. Prospective evaluation of peripheral venous access difficulty in emergency care. Intensive Care Med. 2007 Aug;33(8):1452-7. doi: 10.1007/s00134-007-0634-y. Epub 2007 Jun 7. PMID 17554524
- [Background] Pons PT, Moore EE, Cusick JM, Brunko M, Antuna B, Owens L. Prehospital venous access in an urban paramedic system--a prospective on-scene analysis. J Trauma. 1988 Oct;28(10):1460-3. doi: 10.1097/00005373-198810000-00009. PMID 3172305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We randomly assigned the 26 healthcare providers (16 paramedics, 10 nurses) to use either the BOA® Constricting Band or elastic tourniquets for all IV attempts during the study. Thirteen subjects were in each group. Those that were randomized to the BOA group received training in the use of the device according to the manufacturer's instructions.
Period: Overall Study
Arm/Group | BOA(R) | Standard Care
Started | 243 | 224
Completed | 243 | 224
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BOA(R) | Standard Care | Total
Number analyzed (Participants) | 243 | 224 | 467
Age Categorical [Number; unit: participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 175 | 178 | 353
  >=65 years | 60 | 43 | 103
Age Continuous [Mean (Standard Deviation); unit: years] | 50.17 (19.54) | 46.78 (19.01) | 48.53 (19.34)
Gender [Number; unit: participants]
  Female | 122 | 104 | 226
  Male | 115 | 113 | 228
Region of Enrollment [Number; unit: participants]
  United States | 243 | 224 | 467

OUTCOME MEASURES:

1. Primary Outcome: Success
Description: This outcome will measure self-reported success at starting the peripheral intravenous lines in the upper extremity of adults. Success is defined as an IV line through which blood may be aspirated and flushes freely without evidence of fluid extravasation. To be successful, the IV must be placed within a maximum of three attempts. We will report the number and percentage of patients with successful for both therapies.
Time Frame: five minutes (average)
Measure: Number; unit: participants
Arm/Group | BOA(R) | Standard Care
Number analyzed (Participants) | 243 | 224
participants | 198 | 214

2. Secondary Outcome: First Stick Success
Description: This outcome will report the number of IV attempts as defined by the tip of the needle piercing the skin. The results for each IV attempt will be an ordinal number between one and three. We will compare the number and percentage of patients in each group (1, 2, or 3 sticks) between the two therapies.
Time Frame: Five minutes (average)
Measure: Number; unit: participants
Arm/Group | BOA(R) | Standard Care
Number analyzed (Participants) | 243 | 224
participants | 167 | 186

ADVERSE EVENTS:
Arm/Group | BOA(R) | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/243 | 0/224
Other Adverse Events (participants affected / at risk) | 0/243 | 0/224

LIMITATIONS AND CAVEATS:
There was a significant disparity between subjective opinion and objective results. Nurses and paramedics who used the BOA were uniformly positive in their comments about the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes